CLINICAL TRIAL: NCT02122406
Title: Depression and Anxiety in Rheumatoid Arthritis: Prevalence and Relation With Disease Activity
Brief Title: Depression and Anxiety in Rheumatoid Arthritis
Acronym: DEAR
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Vittorio Grosso, MD, University of Pavia
Other Study IDs: 31748\2009 progetto lorhen
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis; Depression; Anxiety
Keywords: Rheumatoid Arthritis; Depression; Anxiety; DAS28; HADS
MeSH Terms: conditions — Arthritis, Rheumatoid; Depression; Anxiety Disorders | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients RA-BIO: Patients with rheumatoid arthritis treated with biological drugs (infliximab, adalimumab, etanercept, abatacept, tocilizumab, golimumab, certolizumab, rituximab)
  Interventions: Other: Hospital Anxiety and Depression Scale (HADS) questionnaire

INTERVENTIONS:
Other: Hospital Anxiety and Depression Scale (HADS) questionnaire — Patients filled in the Hospital Anxiety and Depression Scale (HADS) questionnaire

SUMMARY:
The primary endpoint of this study is to evaluate the prevalence of anxiety and depressive disorders, and their relationship with disease activity, in patients with rheumatoid arthritis treated with biological drugs

DETAILED DESCRIPTION:
The prevalence of anxiety and depressive disorders will be assesed with the HADS questionnaire at the time of the visit

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* diagnosis of rheumatoid arthritis according to 2010 Classification American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Criteria
* being able to compile questionnaire
* current treatment with biological disease-modifying antirheumatic drug

Exclusion Criteria:

* Current treatment for anxiety or depressive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis currently treated with biological drugs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Caporali, MD, Study Director — University of Pavia
Locations (1):
- IRCCS policlinico San Matteo - Reparto di Reumatologia, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients RA-BIO: Patients with rheumatoid arthritis treated with biological drugs
Period: Overall Study
Arm/Group | Patients RA-BIO
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients RA-BIO
Number analyzed (Participants) | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.35 [54.09 to 76.03]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 29
Region of Enrollment [Number; unit: participants]
  Italy | 200
Disease Duration [Median (Inter-Quartile Range); unit: years] | 11.24 [7.29 to 19.46]
Disease Activity Score on 28 joints (DAS28) [Mean (Standard Deviation); unit: units on a scale] — The Disease Activity Score 28 (DAS28) is a combined index that measures the disease activity in patients with Rheumatoid Arthritis. It is based on the assessment of the number of swollen and tender joints and measure of the ESR.
  Lower values indicate lower disease activity levels. It ranges from 0.49 to 9.35.
  units on a scale | 3.01 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Time Frame: 1 day of enrollement
Measure: Number; unit: participants
Arm/Group | Patients RA-BIO
Number analyzed (Participants) | 200
participants
  HEALTHY | 107
  ANXIETY | 46
  DEPRESSION | 20
  ANXIETY/DEPRESSION | 27

ADVERSE EVENTS:
Time Frame: at the time of the visit
Arm/Group | Patients RA-BIO
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No